CLINICAL TRIAL: NCT01015963
Title: A Study of the Docetaxel Pharmacodynamics and Polymorphisms in ABCC2 and SLC01B3 in Caucasian and African-American Cancer Patients
Brief Title: Studying DNA in Tissue Samples From Caucasian and African-American Cancer Patients Who Received Docetaxel on Clinical Trial CLB-9871
Status: Completed | Type: Observational
Sponsor: Alliance for Clinical Trials in Oncology (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Other Study IDs: CALGB-60805; CALGB-60805; CDR0000617756 (Registry Identifier: NCI Physician Data Query); U10CA031946 (NIH)
Record Dates: First submitted 2009-11-17; First posted 2009-11-18 (Estimated); Last update posted 2017-07-13 (Actual); Status verified 2017-07

CONDITIONS: Bladder Cancer; Breast Cancer; Head and Neck Cancer; Lung Cancer; Unspecified Adult Solid Tumor, Protocol Specific
Keywords: recurrent breast cancer; stage IIIA breast cancer; stage IIIB breast cancer; stage IIIC breast cancer; stage IV breast cancer; extensive stage small cell lung cancer; recurrent small cell lung cancer; recurrent non-small cell lung cancer; stage IIIA non-small cell lung cancer; stage IIIB non-small cell lung cancer; stage IV non-small cell lung cancer; stage IV bladder cancer; recurrent bladder cancer; stage III bladder cancer; recurrent lymphoepithelioma of the nasopharynx; recurrent squamous cell carcinoma of the nasopharynx; stage III lymphoepithelioma of the nasopharynx; stage III squamous cell carcinoma of the nasopharynx; stage IV lymphoepithelioma of the nasopharynx; stage IV squamous cell carcinoma of the nasopharynx; pulmonary carcinoid tumor; recurrent basal cell carcinoma of the lip; recurrent squamous cell carcinoma of the lip and oral cavity; stage III basal cell carcinoma of the lip; stage III squamous cell carcinoma of the lip and oral cavity; stage IV basal cell carcinoma of the lip; stage IV squamous cell carcinoma of the lip and oral cavity; recurrent adenoid cystic carcinoma of the oral cavity; recurrent mucoepidermoid carcinoma of the oral cavity; recurrent verrucous carcinoma of the oral cavity; stage III adenoid cystic carcinoma of the oral cavity; stage III mucoepidermoid carcinoma of the oral cavity; stage III verrucous carcinoma of the oral cavity; stage IV adenoid cystic carcinoma of the oral cavity; stage IV mucoepidermoid carcinoma of the oral cavity; stage IV verrucous carcinoma of the oral cavity; recurrent lymphoepithelioma of the oropharynx; recurrent squamous cell carcinoma of the oropharynx; stage III lymphoepithelioma of the oropharynx; stage III squamous cell carcinoma of the oropharynx; stage IV lymphoepithelioma of the oropharynx; stage IV squamous cell carcinoma of the oropharynx; recurrent squamous cell carcinoma of the hypopharynx; stage III squamous cell carcinoma of the hypopharynx; stage IV squamous cell carcinoma of the hypopharynx; recurrent squamous cell carcinoma of the larynx; recurrent verrucous carcinoma of the larynx; stage III squamous cell carcinoma of the larynx; stage III verrucous carcinoma of the larynx; stage IV squamous cell carcinoma of the larynx; stage IV verrucous carcinoma of the larynx; recurrent esthesioneuroblastoma of the paranasal sinus and nasal cavity; recurrent inverted papilloma of the paranasal sinus and nasal cavity; recurrent midline lethal granuloma of the paranasal sinus and nasal cavity; recurrent squamous cell carcinoma of the paranasal sinus and nasal cavity; stage III esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage III inverted papilloma of the paranasal sinus and nasal cavity; stage III midline lethal granuloma of the paranasal sinus and nasal cavity; stage III squamous cell carcinoma of the paranasal sinus and nasal cavity; stage IV esthesioneuroblastoma of the paranasal sinus and nasal cavity; stage IV inverted papilloma of the paranasal sinus and nasal cavity; stage IV midline lethal granuloma of the paranasal sinus and nasal cavity; stage IV squamous cell carcinoma of the paranasal sinus and nasal cavity; recurrent salivary gland cancer; stage III salivary gland cancer; stage IV salivary gland cancer; recurrent metastatic squamous neck cancer with occult primary; unspecified adult solid tumor, protocol specific; tongue cancer
MeSH Terms: conditions — Urinary Bladder Neoplasms; Breast Neoplasms; Head and Neck Neoplasms; Lung Neoplasms; Small Cell Lung Carcinoma; Carcinoma, Non-Small-Cell Lung; Squamous Cell Carcinoma of Head and Neck; Esthesioneuroblastoma, Olfactory; Salivary Gland Neoplasms; Tongue Neoplasms

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Retrospective
Biospecimen Retention: Samples With DNA — Blood

GROUPS / COHORTS (1):
- Ancillary-correlative (DNA sample analysis): Blood samples collected on clinical trial CLB-9871 are examined via ABCC2 and SLC01B3 genotyping using TaqMan analysis. Other genes related to the pharmacokinetics and side effects of docetaxel may be considered for future genotyping. In some cases, panels of drug response SNPs on high-density arrays may be genotyped.
  Interventions: Other: laboratory biomarker analysis

INTERVENTIONS:
Other: laboratory biomarker analysis — Perform DNA sample analysis

SUMMARY:
This research trial studies deoxyribonucleic acid (DNA) in blood samples from Caucasian and African-American cancer patients who received docetaxel on clinical trial CLB-9871. Studying samples of blood from patients with cancer in the laboratory may help doctors learn more about changes that occur in DNA and identify biomarkers related to cancer. It may also help doctors learn more about how docetaxel is used by the body.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. To determine the genotype of ATP-binding cassette, sub-family C (CFTR/MRP), member 2 (ABCC2) and solute carrier organic anion transporter family, member 1B3 (SLCO1B3) (and other genes potentially relevant in the pharmacokinetics and pharmacodynamics of docetaxel in the future) in Caucasian and African-American cancer patients enrolled on clinical trial CLB-9871.

II. Explore the relationships between these genotypes and docetaxel pharmacokinetic parameters (e.g., area under curve [AUC], steady-state volume of distribution [Vdss]).

OUTLINE:

Blood samples collected on clinical trial CLB-9871 are examined via ABCC2 and SLC01B3 genotyping using TaqMan analysis. Other genes related to the pharmacokinetics and side effects of docetaxel may be considered for future genotyping. In some cases, panels of drug response single nucleotide polymorphisms (SNPs) on high-density arrays may be genotyped.

ELIGIBILITY:
* Registration to CALGB 9871
* Samples present within the CALGB Pathology Coordinating Office that are sufficient to meet study aims

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients enrolled on CLB-9871
Sampling Method: Non-Probability Sample
Enrollment: 69 (Actual)
Dates: Start 2008-10; Primary Completion 2013-01 (Actual); Study Completion 2013-01-01 (Actual)

PRIMARY OUTCOMES:
Incidence of ABBC2 polymorphism (rs12762549) and a SLC01B3 polymorphism (rs11045585) with docetaxel exposure | Up to 2 years
Incidence of SLC01B3 polymorphism (rs11045585) | Up to 2 years

SECONDARY OUTCOMES:
Incidence of grade III/IV leukopenia/neutropenia (induced by docetaxel) | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Lionel D. Lewis, MD, Study Chair — Norris Cotton Cancer Center

REFERENCES:
- [Result] Lewis LD, Miller AA, Owzar K, Bies RR, Markova S, Jiang C, Kroetz DL, Egorin MJ, McLeod HL, Ratain MJ; Alliance for Clinical Trials in Oncology. The relationship of polymorphisms in ABCC2 and SLCO1B3 with docetaxel pharmacokinetics and neutropenia: CALGB 60805 (Alliance). Pharmacogenet Genomics. 2013 Jan;23(1):29-33. doi: 10.1097/FPC.0b013e32835b16d8. PMID 23188068